CLINICAL TRIAL: NCT01124084
Title: The Factors Affecting Intentions of Medical Staff to Use Personal Health Record in Northern Hospitals of Taiwan
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Taipei Medical University (Other)
Responsible Party: Hsyien-Chia Wen, Taipei Medical University Department of Health Care
Other Study IDs: 99014
Record Dates: First submitted 2010-05-11; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Healthy Subjects; Health Care Providers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Health Care Providers

SUMMARY:
Application of health information technology be able to solve a lot of problems of medical management, and effective actions to achieve the purpose of medical care. The "Personal Health Record" (PHR), so that patients can have, access and update their health records and share health information to a new healthcare provider can avoid the duplication of a clinic procedures, reduce medical costs and time, and can make an appointment online, tracking vaccinations, check drug allergy, master with health-related information such as exercise, diet condition, and have no time constraints to the hospital clinic. In the future, PHR is expected to reduce medical errors, reduce costs, effective use of medical resources. Purpose of this study is to understand the impact to the staff's attitude and intention when they use the PHR, and to explore the medical records of personal health awareness and intention to use the relevant factors, the research result will be a reference to government authority or medical institutions in order to promote personal health record system in Taiwan.

In this study, there will include the medical staff of three hospitals in Taipei, the Technology Acceptance Model (TAM model) based structured questionnaire will be used, questionnaire had tested by validity and reliability. The electronic questionnaires will be used, and apply the software SPSS and Amos17.0 descriptive and inferential statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Health care provider
* Volunteer Subject
* Be able to understand the content of questionnaire

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health care providers from three hospitals in Taipei
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hsyien-Chia Wen, Ph.D., Study Chair — Taipei Medical University Department of Health Care
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taipei, Taiwan